CLINICAL TRIAL: NCT00324064
Title: Sexually Dimorphic Effects of GHRH in Adult Growth Hormone Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Mark Clements, Children's Mercy Hospitals and Clinics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06 03-053
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: GHRH/arginine stimulation testing — GHRH(Geref) 1mcg/kg IVP followed by Arginine 10% solution 0.5mg/kg (maximum of 30 Gm) infused over 30 minutes. Labs drawn 6 times over 2 hours.

SUMMARY:
Specific Aim 1 Healthy male and female subjects and growth hormone (GH) deficient subjects display sexually dimorphic GH responses to GHRH administration

Specific Aim 2 GH responses to GHRH in both healthy controls and in GH deficient patients correlate with expression and activity of the stimulatory G proteins, G alpha q and G alpha S. G protein levels correlate with gonadal steroid levels.

Specific Aim 3 Sexually dimorphic GH responses to GHRH are enhanced in Tanner Stage V compared to Tanner Stage 1 individuals

DETAILED DESCRIPTION:
Growth hormone deficiency affects disproportionately more males than females. Although ascertainment bias plays a role in this sexual dimorphism, no plausible mechanism to fully explain this difference has been proposed.

This investigator initiated study will provide currently unavailable data on sexual/age differences in response to GH stimulation testing. Data obtained from the study may provide a basis for developing appropriate normal ranges for adult GH testing, may provide a plausible mechanism for the enhanced hormone responsiveness observed in females, and may provide data on when the sexual differences to GH stimulation may develop.

The objectives of this study are to:

1. Confirm the sexual dimorphism in growth hormone responses for adult growth hormone testing in healthy male and female subjects
2. Correlate peak Growth Hormone Releasing Hormone (GHRH)/arginine induced growth hormone responses with G protein levels in healthy subjects and in patients with a history of childhood GH deficiency
3. Determine whether sexual dimorphism is acquired during puberty

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Males and females, Tanner stage V aged 15-40 years of age with no known endocrine problems
* Males and females, Tanner stage I, aged 5-8 years with no known endocrine problems

GH subjects - Males and females, Tanner stage V, aged 15-21 years with a history of childhood growth hormone deficiency

Exclusion Criteria:

Healthy subjects

* History of GH deficiency or treatment or other known endocrine disorder
* Current height or adult height <5th %
* Female subjects using hormonal methods of birth control
* Female subjects with irregular menstrual cycles

GH subjects

- Subjects with GH deficiency who have not discontinued GH treatment for at least 2 months

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Serum GH levels in response to GHRH/arginine stimulation | End of study

SECONDARY OUTCOMES:
mRNA and protein levels of G alpha q and G alpha S stimulatory proteins | end of study
Serum gonadal steroid levels in the three subject groups | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jill Jacobson, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States